CLINICAL TRIAL: NCT06503484
Title: Utilizing a Brain-Computer Interface for Observational Imitation Training to Enhance Upper Limb Motor Recovery Post-Stroke: A Randomized Controlled Trial
Brief Title: fNIRS-BCI Neurofeedback in Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Hospital, Queen Mary Hospital and University Hospital RWTH Aachen/RWTH Aachen University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20231203001
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Stroke; Brain-computer interface
MeSH Terms: conditions — Stroke | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCI neurofeedback training (Experimental): Patients will perform kinesthetic motor imagery of the affected upper extremity in response to auditory cues from the BCI system. The averaged oxygenated hemoglobin (HbO) level, extracted from optimal channels identified during the localizer session, will serve as signal intensity. This intensity, quantified as percent signal change relative to baseline, will trigger neurofeedback when reaching a predefined threshold. Visual feedback, delivered via the digital mirror therapy system, will guide patients to perform observational imitation tasks using bilateral upper extremities. Each session will include 5-6 movements tailored to the patient's functional performance. After observational imitation training, patients will practice functional adaptation tasks in a virtual environment, where they apply learned movements to functional activities. Sessions will last approximately 75 minutes.
  Interventions: Device: Brain-computer interface
- Sham BCI neurofeedback training (Sham Comparator): In the sham group, patients will wear a similar headset equipment as those in the BCI group. However, the visual feedback provided through the digital mirror therapy system will not be based on their own brain activity. Instead, it will be derived from the brain activity of a participant in the BCI group using the simulation mode of Turbo-Satori. Patients in the sham group will receive constant visual feedback, with a fixed duration of 60 seconds for motor imagery, regardless of their actual brain signals. Like the BCI group, patients will be instructed to use kinesthetic motor imagery and imitate the movement when receiving visual feedback, and practice functional adaptation tasks after observational imitation training. The sham training will also last for around 75 minutes per session.
  Interventions: Device: Sham brain-computer interface

INTERVENTIONS:
Device: Brain-computer interface — Patients will perform kinesthetic motor imagery of the affected upper extremity in response to auditory cues from the BCI system. The averaged oxygenated hemoglobin (HbO) level, extracted from optimal channels identified during the localizer session, will serve as signal intensity. This intensity, quantified as percent signal change relative to baseline, will trigger neurofeedback when reaching a predefined threshold. Visual feedback, delivered via the digital mirror therapy system, will guide patients to perform observational imitation tasks using bilateral upper extremities. Each session will include 5-6 movements tailored to the patient's functional performance. After observational imitation training, patients will practice functional adaptation tasks in a virtual environment, where they apply learned movements to functional activities. Sessions will last approximately 75 minutes.
  Arms: BCI neurofeedback training
Device: Sham brain-computer interface — In the sham group, patients will wear a similar headset equipment as those in the BCI group. However, the visual feedback provided through the digital mirror therapy system will not be based on their own brain activity. Instead, it will be derived from the brain activity of a participant in the BCI group using the simulation mode of Turbo-Satori. Patients in the sham group will receive constant visual feedback, with a fixed duration of 60 seconds for motor imagery, regardless of their actual brain signals. Like the BCI group, patients will be instructed to use kinesthetic motor imagery and imitate the movement when receiving visual feedback, and practice functional adaptation tasks after observational imitation training. The sham training will also last for around 75 minutes per session.
  Arms: Sham BCI neurofeedback training

SUMMARY:
Objectives: 1) To compare the effects of closed-loop brain-computer interface (BCI) driven observational imitation training versus sham BCI open-loop observational imitation training on improving upper limb motor functions in patients with stroke; 2) To investigate whether stroke patients receiving closed-loop training exhibit higher activation levels in the mirror neurons, measured by event-related desynchronization (ERD), compared to those receiving open-loop training.

Hypothesis to be tested: The closed-loop training is more effective than open-loop training in improving upper limb motor outcomes, and there is an increase in the mirror neurons activity in those receiving closed-loop training.

Design and subjects: A randomized controlled trial with 44 participants with stroke.

Study instruments: Functional near-infrared spectroscopy (fNIRS)-based BCI and electroencephalography (EEG).

Interventions: In the BCI training, participants will engage in kinesthetic motor imagery. When the M1 activation level recorded by fNIRS surpasses a predefined threshold, participants will receive visual feedback to guide them to imitate the movement. However, for participants in the sham BCI group, the visual feedback will be given will be given constantly. Both types of training consist of ten sessions.

Main outcome measures: Upper limb motor tests and the activity of mirror neurons measured by sensorimotor ERD using EEG.

Data analysis: Analysis of variance and correlation. Expected results: The closed-loop BCI-driven observational imitation training is more effective than sham BCI open-loop training on enhancing hemiplegic upper limb functions and the activation of the mirror neurons in patients after stroke.

DETAILED DESCRIPTION:
Objectives: 1) To compare the effects of closed-loop brain-computer interface (BCI) driven observational imitation training versus sham BCI open-loop observational imitation training on improving upper limb motor functions in patients with stroke; 2) To investigate whether stroke patients receiving closed-loop training exhibit higher activation levels in the mirror neurons, measured by event-related desynchronization (ERD), compared to those receiving open-loop training.

Hypothesis to be tested: The closed-loop training is more effective than open-loop training in improving upper limb motor outcomes, and there is an increase in the mirror neurons activity in those receiving closed-loop training.

Design and subjects: A randomized controlled trial with 44 participants with stroke.

Study instruments: Functional near-infrared spectroscopy (fNIRS)-based BCI and electroencephalography (EEG).

Interventions: In the BCI training, participants will engage in kinesthetic motor imagery. When the M1 activation level recorded by fNIRS surpasses a predefined threshold, participants will receive visual feedback to guide them to imitate the movement. However, for participants in the sham BCI group, the visual feedback will be given constantly. Both types of training consist of ten sessions.

Main outcome measures: Upper limb motor tests and the activity of mirror neurons measured by sensorimotor ERD using EEG.

Data analysis: Analysis of variance and correlation. Expected results: The closed-loop BCI-driven observational imitation training is more effective than sham BCI open-loop training on enhancing hemiplegic upper limb functions and the activation of the mirror neurons in patients after stroke.

ELIGIBILITY:
Inclusion Criteria

1. unilateral upper extremity motor deficits caused by ischemic stroke, confirmed by medical documents such as discharge summary and/or neuroimaging examinations.
2. chronic phase of stroke, i.e., time after stroke onset more than six months.
3. aged between 18 and 75 years old.
4. with mildly-to-moderately impaired upper limb functional activity that is stratified according to the levels 3-7 in the Functional Test for the Hemiplegic Upper Extremity.
5. able to give informed written consent to participate in the study.
6. able to read and understand traditional Chinese.

Exclusion Criteria

1. previous diagnosis of any neurological disease excluding ischemic stroke.
2. presence of any sign of cognitive problems (The Montreal cognitive assessment Hong Kong version<22/30).
3. Severe spasticity measured by the Modified Ashworth Scale score>2 in the hand, wrist or elbow extensor muscle in the hemiparetic upper extremity.
4. with other notable impairments of the upper limb not caused by stroke (e.g., bone fracture in the past year, congenital deformity, or other impairments).
5. current participation in any other treatment programme or clinical study involving exercise, non-invasive brain stimulation, or BCI/neurofeedback.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) | Baseline
  The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) evaluates upper limb motor impairment post-stroke. It assesses the movement, coordination, and reflex actions of the hemiplegic upper limb. The total scores are 66.
The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) | At 2 weeks
  The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) evaluates upper limb motor impairment post-stroke. It assesses the movement, coordination, and reflex actions of the hemiplegic upper limb. The total scores are 66.
The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) | At one-month
  The Fugl-Meyer Assessment - Upper Extremity Scores (FMA-UE) evaluates upper limb motor impairment post-stroke. It assesses the movement, coordination, and reflex actions of the hemiplegic upper limb. The total scores are 66.

SECONDARY OUTCOMES:
The Action Research Arm Test (ARAT) | Baseline
  The Action Research Arm Test (ARAT) is an assessment for upper limb functional activities post-stroke, with four subscales to evaluate grasp, grip, pinch, and gross movement, with total scores of 57.
The Action Research Arm Test (ARAT) | At 2 weeks
  The Action Research Arm Test (ARAT) is an assessment for upper limb functional activities post-stroke, with four subscales to evaluate grasp, grip, pinch, and gross movement, with total scores of 57.
The Action Research Arm Test (ARAT) | At one-month
  The Action Research Arm Test (ARAT) is an assessment for upper limb functional activities post-stroke, with four subscales to evaluate grasp, grip, pinch, and gross movement, with total scores of 57.

CONTACTS AND LOCATIONS:
Locations (1):
- Jack Jiaqi Zhang, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided